CLINICAL TRIAL: NCT02858882
Title: Vitamin D Status and Muscle Function Among Adolescent and Young Swimmers.
Brief Title: Vitamin D Status and Muscle Function
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Team Denmark (Other); Hvidovre University Hospital (Other); Danmarks Fødevareforskning (Unknown); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Other Study IDs: KF01322182
Record Dates: First submitted 2016-07-27; First posted 2016-08-08 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Vitamin D Status; Muscle Function
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Swimmers: Screening of elite athletes
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Screening of elite swimmers

SUMMARY:
People living at Northern latitudes are at risk of suffering from vitamin D insufficiency due to low sun exposure and the risk may be even more pronounced among elite swimmers since indoor training further reduces sun exposure. In light of this, the investigators want to examine vitamin D status in young elite swimmers and if there is an association between vitamin D status and muscle strength.

DETAILED DESCRIPTION:
To examine vitamin D status in young elite swimmers and if there is an association between vitamin D status and muscle strength, twenty-nine swimmers, 12 female and 17 male (16-24 years) residing at latitude 55-56°N were included to the trial conducted in March-April. Blood samples were analysed for serum 25-hydroxyvitamin D (s-25(OH)D) and hand-grip strength was measured as marker of muscle strength. Subjects´ vitamin D and calcium intake were assessed by food frequency questionnaire and sun exposure and training status by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Age: 16-35 years

Top atlets, conducting:

* Hard physical activity
* Indoor elitesport min. 10 hours a week
* Healthy, without use of any medications
* Eat fish max 2 times per week

Exclusion Criteria:

* Use of corticosteroids
* Illness
* Use of supplements
* Use of solarium
* Donation of blood within the last 3 months
* Having spent time below the latitude of 42° north from September through April

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2007-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D (s-25(OH)D) | 2 months

SECONDARY OUTCOMES:
Food frequency questionnaire | One week
Hand-grip strength | 2 months

IPD SHARING:
Plan to Share IPD: No